CLINICAL TRIAL: NCT03434548
Title: Longitudinal Adaptive Study of Molecular Pathology and Neuronal Networks in Huntington's Disease Gene-Expansion Carriers (HDGEC) and Healthy Controls Using Positron Emission Tomography (PET) and Multi-modal Magnetic Resonance Imaging (MRI)
Brief Title: IMarkHD: in Vivo Longitudinal Imaging of HD Pathology
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 242859
Record Dates: First submitted 2018-02-07; First posted 2018-02-15 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Huntington Disease
Keywords: Huntington's disease; PET imaging; MRI imaging
MeSH Terms: conditions — Huntington Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Analysis will be performed to confirm the size of the CAG expansion mutation within the HD gene for all PwHD, for research purposes only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Healthy controls. Multi-modal MRI imaging.
  Interventions: Other: Multi-modal MRI imaging
- Cohort 2: People with Huntington's (without symptoms, early disease stage, and later disease stage), and healthy controls
  People with HD divided in groups according to disease stage:
  * Without symptoms (approximately HD-ISS stage 0 or 1)
  * Early disease (approximately HD-ISS stage 2)
  * Later disease stage (approximately HD-ISS stage 3)
  Interventions: Radiation: PET imaging; Other: Multi-modal MRI imaging

INTERVENTIONS:
Radiation: PET imaging — PET imaging Radiation: Radioligand [¹¹C]MePPEP Intravenous injection of radioligand in the arm with PET imaging of the brain. Radiation: Radioligand [¹¹C]IMA107 Intravenous injection of radioligand in the arm with PET imaging of the brain. Radiation: Radioligand [¹¹C]MDL100907 Intravenous injection of radioligand in the arm with PET imaging of the brain. Radiation: Radioligand [¹¹C]MDL100907 Intravenous injection of radioligand in the arm with PET imaging of the brain.
  PET imaging Radiation: Radioligand [¹¹C]MePPEP Intravenous injection of radioligand in the arm with PET imaging of the brain. Radiation: Radioligand [¹¹C]IMA107 Intravenous injection of radioligand in the arm with PET imaging of the brain. Radiation: Radioligand [¹¹C]MDL100907 Intravenous injection of radioligand in the arm with PET imaging of the brain. Radiation: Radioligand [¹¹C]MDL100907 Intravenous injection of radioligand in the arm with PET imaging of the brain.
  Groups: Cohort 2
Other: Multi-modal MRI imaging — Multi-modal MRI imaging

SUMMARY:
iMarkHD is an adaptive, longitudinal positron emission tomography (PET) and magnetic resonance (MR) imaging study in Huntington's disease (HD) that aims to assess abnormal molecular, functional, and structural changes in participants' brains, ranging from several years before symptom onset to the advanced symptom stage. The study will be conducted over a three (3) year period (Baseline, Year-1, and Year-2).

DETAILED DESCRIPTION:
It is likely that, over time, multiple pathophysiological changes influence Huntington's disease (HD) progression. Rather than focusing on one element, the combined PET and multi-modal MRI assessments in this study will allow comprehensive examination of the molecular, functional, and structural framework of HD progression in the brain. The investigators will compare PET and MRI measurements at different disease stages with age- and sex-matched healthy control (HC) participants and monitor, over follow-up visits, to evaluate how specific or combinatorial changes may influence the development of symptoms and disease progression. Furthermore, disease progression markers may be identified that can characterize and predict events preceding symptom development, which could be used as outcome measures in future clinical trials. Study results could also lead to the development of new targeted therapies.

The study has two main objectives. First, to use a series of PET scans to investigate four target receptors in specific areas of the brain that are affected by HD and are thought to be responsible for the motor, cognitive, and behavioral symptoms. Second, to investigate structural and functional changes, including alterations in brain connections, using a multi-modal MRI protocol. The investigators will combine MRI and PET findings with clinical measures to precisely characterize univariate and multivariate markers of disease progression.

There will be two (2) cohorts in this study. Cohort 1 will consist of five (5) HC participants (who do not have the HD gene mutation) recruited and enrolled to enable optimization of MRI imaging techniques. Each participant in Cohort 1 will complete a minimum of 3 visits. Cohort 2 will consist of 72 people with HD (PwHD) and 36 HC participants; each participant will complete a minimum of 10 visits over three (3) years. The 72 PwHDs will be recruited into three (3) groups depending on disease stage: 24 PwHDs who do not have symptoms and are predicted to develop clinically relevant symptoms in a few years; 24 PwHDs with symptoms in early disease stages; and 24 PwHDs with symptoms in advanced disease stages.

The investigators will conduct a preliminary analysis after all baseline visits are completed and a decision will be made whether to add an additional group of 24 PwHDs with no symptoms and who are several years away from developing symptoms, and an additional 12 HCs. After 50% of participants have completed Year 2 follow-up visits, preliminary analysis will be carried out to determine whether to extend the study to include a Year 3 follow-up visit which would be identical to the Year 1 and 2 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

PwHDs and HC participants:

* Female and male adults, aged 21-75 years old, inclusive.
* Adequate visual (Snellen chart) and auditory (Rinne and Weber tests) acuity to complete the psychological testing as determined by the investigator.
* Capable of giving informed consent.
* Willing to comply with highly effective contraceptive measures following informed consent (for Cohort 2 only).
* Vital signs within certain set ranges.
* Considered by the investigator to be in good health as judged by the absence of clinically significant diseases, laboratory values, physical examination, and able to travel to imaging and clinical assessment centers in London, UK.
* Suitable physically and psychologically to travel (with a companion if requested) and undergo the assessments as judged by the investigator.

PwHDs without symptoms: (approximately HD-ISS stage 0 or 1)

* HDGECs with ≥ 40 CAG repeats
* TMS ≤ 6 AND TFC ≥ 12 AND CAP > 70 PwHDs with symptoms in early disease: (approximately HD-ISS stage 2)
* HDGECs with ≥ 40 CAG repeats
* If one of the following criteria is met:

  1. TMS ≤ 6 AND TFC = 11
  2. TMS is between 7 and 23 inclusive AND TFC is between 11 and 13 inclusive
  3. TMS is between 24 and 33 inclusive AND SDMT > 50 AND TFC is between 11 and 13 inclusive PwHDs with symptoms in late disease (approximately HD-ISS stage 3)
* HDGECs with ≥ 40 CAG repeats
* If one of the following criteria is met:

  1. TMS ≤ 6 AND TFC is between 7 and 10 inclusive
  2. TMS is between 7 and 23 inclusive AND TFC is between 8 and 10 inclusive
  3. TMS is between 24 and 33 inclusive AND SDMT > 50 AND TFC is between 7 and 10 inclusive
  4. TMS is between 7 and 23 inclusive AND TFC = 7
  5. TMS > 23 AND SDMT ≤ 50 AND TFC is between 7 and 13 inclusive
  6. TMS > 33 AND SDMT > 50 AND TFC is between 7 and 13 inclusive

Healthy Controls (HC):

* Age- and sex-matched, and balanced (±8 years) with PwHDs.
* No known family history of HD or have known family history of HD but have been tested for the huntingtin gene glutamine codon (CAG) expansion and are not at genetic risk for HD (CAG < 36).

Exclusion Criteria:

PwHD and HC participants:

* Presence or history of other neurological condition (including brain surgery, intracranial hematoma, stroke/cerebrovascular disorders, demyelinating conditions, epilepsy) likely to interfere with imaging or PET studies or abnormal neurologic examination finding suggestive of a central nervous system pathology (for PwHDs - other than HD).
* Presence or history of primary psychiatric disorders unrelated to HD.
* Participants using any medications with known actions on cannabinoid type 1 receptors (CB1R), phosphodiesterase 10A (PDE-10A), 5-hydroxytryptamine-2A receptor (5-HT2AR), histamine type-3 receptors (H3R), or any other PET targets used in iMarkHD.
* Pregnancy confirmed by a positive urine pregnancy test.
* Participants who are currently breastfeeding or intend to breastfeed during the study.
* Contraindication to MRI, such as presence of metal devices or implants (e.g. pacemaker, vascular- or heart- valves, stents, clips), metal deposited in the body (e.g. bullets or shells), or metal grains in the eyes.
* History of alcoholism or substance abuse within 3 years prior to study entry.
* Failure of drug screen for substances of abuse such as amphetamines, barbiturates, benzodiazepines, methadone, opiates, cocaine, cannabinoids, phencyclidine, and creatine.
* History of cancer.
* Claustrophobia.
* Significant back pain that makes prolonged laying on the PET or MRI scanner intolerable.
* Contraindication for arterial cannulation as judged by the Allen test and the laboratory blood screening for coagulopathy (Cohort 2 only).
* Inability to communicate or cooperate with the principal investigator/iMarkHD team for any reason.
* Participants who are currently enrolled in or participated in clinical trials testing the efficacy of novel therapeutics with action on the specific PET targets being tested within 3 months of screening.
* Any concurrent conditions that could interfere with the safety and/or tolerability measurements.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with Huntington's disease (PwHD) and healthy controls (HCs). PwHD participants will be recruited from specialty clinics known as Participant Identification Centers (Human Genetics, Neurology, Psychiatry) that advise and treat people affected by HD. Participants may receive information about the study through a website, clinical practices, advocacy newsletters, or other approved sources. Community controls will be recruited using advertisements, flyers, and newsletters with the support of the iMarkHD operational staff.
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure 1 | 2 years
  Quantitative change in binding profile of four discrete molecular PET markers over the period of 2 years.
  These markers include:
  1. Cannabinoid 1 Receptor binding.
  2. Phosphodiesterase 10A enzyme binding.
  3. 5-hydroxytryptamine-2A receptor binding.
  4. Histamine type-3 receptor binding.
  The study will assess basal ganglia and cortical pathology with four highly specific PET radioligands ([11C]MePPEP, [11C]IMA107, [11C]MDL100907 and [11C]MK-8278), tagging 4 targets of interest: cannabinoid type 1 receptors (CB1R), phosphodiesterase 10A (PDE-10A), 5-hydroxytryptamine-2A receptor (5-HT2AR) and histamine type-3 receptors (H3R), respectively, at baseline, 1 and 2years. The main focus will be on the basal ganglia.
Primary outcome measure 2 | 2 years
  Determine whether selected PET markers could be used as markers of HD disease progression and treatment response in therapeutic trials.
  These markers include:
  1. Cannabinoid 1 Receptor binding.
  2. Phosphodiesterase 10A enzyme binding.
  3. 5-hydroxytryptamine-2A receptor binding.
  4. Histamine type-3 receptor binding.
  The study will assess basal ganglia and cortical pathology with four highly specific PET radioligands ([11C]MePPEP, [11C]IMA107, [11C]MDL100907 and [11C]MK-8278), tagging 4 targets of interest: cannabinoid type 1 receptors (CB1R), phosphodiesterase 10A (PDE-10A), 5-hydroxytryptamine-2A receptor (5-HT2AR) and histamine type-3 receptors (H3R), respectively, at baseline, 1 and 2years. These outcomes will be linked to scale-based and other clinical outcomes performed over the same timelines to determine the link between clinically defined disease progression and the PET markers.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Williams, PhD, Study Chair — King's College London; Daniel J van Wamelen, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided